CLINICAL TRIAL: NCT00417365
Title: "A Comparison Study of the WaterWorks® Douching Device vs. Commercial OTC Douching Device for the Reduction or Abatement of Perceived Vaginal Odor With or Without Complaints of Discharge in Women With no Infectious Causes of Vaginitis"
Brief Title: Efficacy of (WaterWorks®)Douching Device for Elimination of Perceived Vaginal Odor Not Caused by BV or Vaginitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abbott Research Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARG105B; Pre-IDE I060071
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-08

CONDITIONS: Vaginal Odor
Keywords: odor; douching; BV; vaginitis; vaginal; yeast; ecosystem; Lactobacilli; Nugent; Amsel
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Who Masked: Investigator

INTERVENTIONS:
Device: WaterWorks Douching Device

SUMMARY:
Comparing the new Stainless Steel WaterWorks® douching device to a commercially available douching device using just water for safety and efficacy of odor abatement.

DETAILED DESCRIPTION:
Vaginal symptoms, including abnormal odor with or without complaints of discharge, are relatively common complaints. It is generally assumed that most women with these complaints have a vaginal infection, bacterial vaginosis, trichomoniasis, or vulvovaginal candidiasis. However, investigators suggest that there is a large population of women who complain of odor with or without complaints of discharge, and in whom no clear cause can be found. For these women, there are currently no treatment options.

Anecdotal evidence suggests that stainless steel used with just water has an effect in reducing odors and is so used to reduce odors on hands by chefs. The Water Works® Douching Device is a light-weight (1oz) stainless steel douching device that was developed to aid in the treatment of vaginal odor. Additional anecdotal evidence suggests that douching with the Water Works® Douching Device had little or no affect on the vaginal Eco-System (e.g. good bacteria, Lactobacilli).

This study (ARG105B) will compare the Water Works® Douching Device to a commercially available over the counter douching device for the ability to reduce or eliminate abnormal odor (with or without complaints of discharge) in women with this subjective complaint, but no objective findings of a vaginal infection. The study will also compare the Water Works® Douching Device to the commercial device with respect to the adverse effect of the vaginal Eco-System.

ELIGIBILITY:
Inclusion Criteria:

Enrollment in the study will be open to those subjects who meet the following inclusion criteria:

1. Non-pregnant females, 18 years and older
2. Complaint of abnormal vaginal odor with or without complaints of discharge
3. Subject with perceived, abnormal vaginal odor on the date she is evaluated
4. Odor scale 4 cm or greater (using the subject's perception visual analog rating scale of 10 cm): 0 = no odor 10 = strong offensive odor
5. Subject is not fulfilling Amsel's criteria for BV listed below (only meets 0 or 1 Amsel's criteria)
6. Not treated for Bacterial Vaginosis, VVC, intra-vaginal or oral anti-fungal medications or antibiotics, within the last 14 days of enrollment
7. Willing and able to comply with study requirements
8. Has provided written informed consent

Exclusion Criteria:

Subjects will be excluded from the enrollment if they have any of the following:

1. Odor scale less than 4 cm (on the Visual Analog rating scale of 10 cm)
2. Subjects with presence of BV
3. Subjects with other lower genital tract infections (e.g., symptomatic VVC, trichomoniasis, Chlamydia trachomatis, Neisseria gonorrhoeae or herpes simplex virus)
4. Subjects with another vaginal or vulvar condition, which would confound the interpretation of clinical response
5. Subjects who received antifungal or antimicrobial therapy (systemic or intravaginal) within the last 14 days
6. Subjects who will be under treatment during the study period for cervical intra-epithelial neoplasia (CIN) or cervical carcinoma
7. Positive pregnancy test
8. Any abnormal anatomy or pathology of the subject's vagina
9. Known HIV positive
10. Pap smear >LSIL (untreated or not evaluated) [LSIL = Low-grade squamous intraepithelial lesion]
11. Subject currently having a menstrual period (excluded until completion of period)
12. Subjects with a body mass index (BMI) of 39 or greater
13. Investigator believes that external factor(s) is producing odor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-08; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is the reduction or abatement of the
subject's perceived vaginal odor as determined at Visit 3.
This improvement will be measured using a visual analog scale that
asks subjects to rate their perception of vaginal odor on a scale that
is anchored at two extremes, "no odor", and, "strong offensive odor".

SECONDARY OUTCOMES:
Effects on the vaginal Eco-System will be assessed using the
Lactobacilli score and the Nugent score. The safety profile of the douching
device (Water Works® versus control) will be assessed through the collection
of any reported adverse events. Any adverse event, will be reported in terms
of severity, relationship to treatment, duration, and resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Chatwani, M.D., Principal Investigator — Temple University; Jack Sobel, M.D., Principal Investigator — Wayne State University
Locations (7):
- United States (7):
  - Segal Institute of Clinical Research, Aventura, Florida
  - Discovery Research, Inc., Plantation, Florida
  - Atlanta Women's Research Institute, Atlanta, Georgia
  - Wayne State University, Harper Hospital, Detroit, Michigan
  - Salem Research, Winston-Salem, North Carolina
  - University of Oklahoma, Tulsa, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Infectious Diseases in Obstetrics and Gynecology Volume 2006 (2006), Article ID 95618, 4 pages doi:10.1155/IDOG/2006/95618 /Published results are from ARG sponsored study ARG105.
- [Derived] Hassan S, Chatwani A, Brovender H, Zane R, Valaoras T, Sobel JD. Douching for perceived vaginal odor with no infectious cause of vaginitis: a randomized controlled trial. J Low Genit Tract Dis. 2011 Apr;15(2):128-33. doi: 10.1097/LGT.0b013e3181fb4270. PMID 21263351